CLINICAL TRIAL: NCT07010224
Title: Clinical Characteristics of Elastofibroma Dorsi, Long-Term Outcomes After Surgical Resection, and Analysis of Risk Factors
Brief Title: Elastofibroma Dorsi: Clinical Features, Surgical Outcomes, and Risk Factors
Status: Active, not recruiting | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Caner İşevi, MD, Dr. Caner İşevi, Thoracic Surgeon, Department of Thoracic Surgery, Ondokuz Mayıs University, Ondokuz Mayıs University
Other Study IDs: B.30.2.ODM.0.20.08/280
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-05

CONDITIONS: Elastofibroma Dorsi
Keywords: Elastofibroma Dorsi; Subscapular Mass; Chest Wall Tumor; Risk Factors; Thoracic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgically Treated Elastofibroma Dorsi Patients: This cohort includes patients diagnosed with elastofibroma dorsi who underwent surgical resection between 2010 and 2025. Patients were retrospectively evaluated for demographic characteristics, clinical features, diagnostic methods, surgical findings, postoperative complications, and recurrence during follow-up.
  Interventions: Other: Retrospective Medical Record Review

INTERVENTIONS:
Other: Retrospective Medical Record Review — Review of archived medical, surgical, and radiological records of patients diagnosed with elastofibroma dorsi and treated surgically. No active intervention was administered as part of the study.

SUMMARY:
This study aims to retrospectively evaluate patients who underwent surgical treatment for elastofibroma dorsi, a rare benign tumor typically located in the subscapular region of the chest wall. The study will analyze demographic and clinical features, risk factors, diagnostic imaging methods, postoperative complications, and recurrence rates. By identifying potential predictors of complications and recurrence, the study hopes to contribute to the understanding and management of this silent and often incidental lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent surgical treatment for elastofibroma dorsi
* Histopathological confirmation of the diagnosis
* Minimum of 1-month postoperative follow-up available
* Age 18 years or older
* Accessible medical and imaging records in hospital archives
* Signed informed consent available in patient records (if applicable)

Exclusion Criteria:

* Patients diagnosed with elastofibroma dorsi but not treated surgically
* Cases without histopathological confirmation
* Incomplete or insufficient medical and radiological records
* Postoperative follow-up period less than 1 month
* Patients younger than 18 years
* Absence of documented informed consent (if applicable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients (aged 18 and older) who were diagnosed with elastofibroma dorsi and underwent surgical resection at a single tertiary care center between 2010 and 2025. All included patients had histopathologically confirmed diagnoses and at least one month of postoperative follow-up available in hospital records.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Completion of Retrospective Data Collection Form | Within 3 months after data collection begins
  Completion of data collection from medical records of patients diagnosed with elastofibroma dorsi who underwent surgical treatment, including demographic features, clinical presentation, imaging modalities, surgical outcomes, postoperative complications, and recurrence.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Nishio J, Isayama T, Iwasaki H, Naito M. Elastofibroma dorsi: diagnostic and therapeutic algorithm. J Shoulder Elbow Surg. 2012 Jan;21(1):77-81. doi: 10.1016/j.jse.2011.01.043. Epub 2011 Apr 27. PMID 21524925